CLINICAL TRIAL: NCT02875938
Title: Effect of Music on Reading Comprehension for Patients With Aphasia
Acronym: EMRA1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CarilionClinic
Record Dates: First submitted 2016-08-10; First posted 2016-08-23 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Aphasia
Keywords: left middle cerebral artery; cerebrovascular accident (CVA); stroke
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Music and reading lyrics (Experimental): A single-subject adapted alternating treatment design will be used to compare two music conditions, using music with sung lyrics simultaneously with silent reading of the lyrics, and priming with music and sung lyrics followed by reading of the lyrics, with a control condition using reading materials without music.
  Interventions: Behavioral: Simultaneous music and reading lyrics; Behavioral: Priming with music; Behavioral: Control

INTERVENTIONS:
Behavioral: Simultaneous music and reading lyrics — music with sung lyrics simultaneously with silent reading of the lyrics.
Behavioral: Priming with music — priming with music and sung lyrics followed by reading of the lyrics.
Behavioral: Control — control condition using reading materials without music.

SUMMARY:
This investigation uses a single-subject, adapted alternating research design to compare two different experimental conditions using music with lyrics combined with visual stimulation of the written lyrics, to extend the emotional word effect to phrases, in order to stimulate reading comprehension of the trained material for patients with aphasia. The two music conditions include 1) music with sung lyrics simultaneously with silent reading of the written lyrics; and 2) music with sung lyrics, followed by silent reading of the written lyrics (i.e. priming with the music). A control set without music will be used additionally within every third session to detect potential history and maturation effects. All conditions will be followed by a silent reading phrase-completion task composed of written words from the total combined sets of stimuli.

DETAILED DESCRIPTION:
The purpose of this investigation is to examine the evidence on emotion, language, and music, and propose a first step, in the form of a single-subject research design, to determine the most effective and efficient method for application to the rehabilitation of patients with aphasia. A single-subject adapted alternating treatment design will be used to compare two music conditions, using music with sung lyrics simultaneously with silent reading of the lyrics, and priming with music and sung lyrics followed by reading of the lyrics, with a control condition using reading materials without music. Risks are expected to be minimal. The risk is confidentiality. Risk management procedures in this study include: assuring confidentiality of participants, assuring qualified personnel, assuring convenient location, ensuring adequate enrollment, continual monitoring, addressing potential conflicts of interest, and making a plan to manage problems. Continual monitoring will be used to assess whether study interventions appear to be interfering with normal speech therapy treatment. If the researcher sees any signs of interference, the subject will be withdrawn from the research and study interventions will be stopped.

ELIGIBILITY:
Inclusion Criteria:

* Post-hospitalization;
* premorbid reading at the 8th grade level or higher based on the participant's/family's stated years of formal education;
* post-stroke aphasia/left middle cerebral artery (MCA) CVA based on electronic medical record (EMR) and computed tomography (CT)/magnetic resonance imaging (MRI) imaging reports, or consult with the neurologist;
* intact left amygdala and left extrastriate cortex based on EMR and CT/MRI imaging reports, or consult with the neurologist;
* reliability in answering yes/no questions as determined by a 90% score on yes/no comprehension therapy tasks during regular speech therapy.

Capacity to provide informed consent concerning a study involving an intervention with music therapy: determined by the physician who refers the patient.

Exclusion Criteria:

* Co-morbidities diagnosed and reported in the EMR or shown on CT scan or MRI including past history of stroke with residual symptoms, dementia, Parkinson's disease, head injury, etc.;
* hemianopsia or other visual field defects affecting vision for reading, and in particular right homonymous hemi- or inferior quadrantanopsia;
* previous history of learning disabilities in reading/writing;
* significant psychiatric diagnosis;
* English as a Second Language or non-English language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Percent correct responses per day on phrase completion task. | through study completion, an average of 1 year
  Differential response to the interventions (counted as the percent correct responses per day.
Number of sessions required to achieve mastery. | through study completion, an average of 1 year
  count number of sessions.
Retention of the reading material | 3 weeks post-intervention.
  Number of items recalled.

SECONDARY OUTCOMES:
International Classification of Functioning, Disability, and Health (ICF) Body Functions/Structures, Activities, and Participation | through study completion, an average of 1 year
  Pretest/post-test information on the ICF Body Functions/Structures, Activities, and Participation (Hurkmans et al. 2011).
Boston Diagnostic Aphasia Examination-Third Edition (BDAE-3) | through study completion, an average of 1 year
  The Boston Diagnostic Aphasia Examination-Third Edition (BDAE-3) (Goodglass, Harold, & Barresi, Austin: PRO-Ed.): Pretest reading scores on the BDAE full version subtests, i.e. B. Word Identification: 1. Word-Picture Match, and 2. Lexical Decision; C. 1. Homophone Matching; D. Derivational and Grammatical Morphology: 1. Matching to spoken sample; E. Oral Reading: 1. Basic oral word reading; F. Oral Reading of Sentences with Comprehension; and G. Reading Comprehension-Sentences and Paragraphs; will be completed prior to baseline A and initiating intervention, and immediately following completion of intervention to assess generalization to non-trained stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline A. Treichler, MS, CCC-SLP, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Franklin Memorial Hospital, Rocky Mount, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT02875938/Prot_SAP_000.pdf